CLINICAL TRIAL: NCT05468502
Title: An Open Clinical Study to Explore the Safety, Tolerance and Preliminary Efficacy of Human Umbilical Cord Mesenchymal Stem Cell Injection in the Treatment of Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Phase I/IIa Clinical Trial of Human Umbilical Cord Mesenchymal Stem Cell Injection in the Treatment of Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Life Science & Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHLF-MSC-101
Record Dates: First submitted 2022-07-12; First posted 2022-07-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Four different doses were set, and three subjects in each dose plan received human umbilical cord mesenchymal stem cell injection successively. Each subject received a single dose of 6.0*10^6, 3.0*10^7, 6.0*10^7, and 1.2*10^8 cells / person.
  Interventions: Drug: Human umbilical cord mesenchymal stem cell injection

INTERVENTIONS:
Drug: Human umbilical cord mesenchymal stem cell injection — Different doses of human umbilical cord mesenchymal stem cell injection were infused to the focus of patients with idiopathic pulmonary fibrosis through bronchoscope, and the tolerance of subjects to different doses of human umbilical cord mesenchymal stem cell injection was observed, and the curative effect was preliminarily observed.

SUMMARY:
Main purpose

-To explore the safety and tolerance of human umbilical cord mesenchymal stem cells in the treatment of idiopathic pulmonary fibrosis (IPF).

Secondary purpose

* To explore the preliminary efficacy of human umbilical cord mesenchymal stem cells in the treatment of idiopathic pulmonary fibrosis (IPF), and to recommend the appropriate dose of cell therapy for subsequent clinical studies.
* To explore the immunogenicity of human umbilical cord mesenchymal stem cell injection in the treatment of idiopathic pulmonary fibrosis (IPF).

This study adopts a clinical research design of multi center, single dose and increasing dose.

18 qualified IPF subjects will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years (inclusive), regardless of gender;
2. Diagnosed with idiopathic pulmonary fibrosis (IPF) according to the 2018 diagnostic guidelines jointly issued by the American Thoracic Society (ATS), European Respiratory Society (ERS), Japanese Respiratory Society (JRS), and Latin American Thoracic Association (ALAT);
3. Subjects with typical HRCT imaging manifestations of IPF (honeycombing, traction bronchiectasis or bronchiolectasis (mainly appearing in ground-glass opacities and fine reticular opacities)) within 12 months prior to screening;
4. Subjects whose disease is assessed by the investigator as stable within 3 months prior to dosing, with diffusing capacity for carbon monoxide (DLCO) at 30%-79% of the predicted value (adjusted for Hb), and FVC/predicted value ≥50%;
5. Blood biochemical tests must meet the following criteria: alanine aminotransferase (ALT) ≤1.5×ULN, aspartate aminotransferase (AST) ≤1.5×ULN, total bilirubin (TBIL) ≤1.5×ULN, direct bilirubin (DBIL) ≤1.5×ULN, serum creatinine (Cr) ≤1.5×ULN;
6. Expected survival ≥12 months;
7. Subjects with good compliance, who are able to understand and cooperate in performing pulmonary function tests, and are willing to receive medication as required by the protocol and undergo follow-up examinations on schedule;
8. Subjects who voluntarily participate in the trial, understand, and sign the informed consent form.

Exclusion Criteria:

1. Subjects, who have previously received stem cell therapy, are intolerant to cell therapy, or have taken drugs that may cause or exacerbate pulmonary fibrosis (such as amiodarone, bleomycin, or methotrexate, etc.);
2. Subjects with interstitial lung disease (ILD) other than IPF, including but not limited to: any other type of interstitial pneumonia; lung diseases associated with exposure to fibrogenic agents or other environmental toxins or drugs; other types of occupational lung diseases; granulomatous lung diseases; pulmonary vascular diseases; systemic diseases, including vasculitis, infectious diseases (i.e., tuberculosis), and connective tissue diseases;
3. Subjects currently requiring oxygen therapy (oxygen therapy time ≥15 hours/day);
4. Subjects with a history of mechanical ventilation or concurrent infectious pneumonia or asthma within 1 month prior to screening;
5. Subjects with a history of malignancy within 5 years prior to screening;
6. Subjects who have been hospitalized three or more times due to acute exacerbation of IPF or other respiratory diseases within 1 year prior to screening;
7. Evidence of current digestive, urinary, cardiovascular, cerebrovascular, hematological, neurological, psychiatric, or metabolic diseases that may affect safety, such as poorly controlled type 2 diabetes (fasting blood glucose ≥10.0 mmol/L or HbA1c ≥8.5%) or poorly controlled hypertension (≥160/100 mmHg).
8. History of psychotropic drug abuse or drug addiction;
9. Known history of immune system diseases (e.g., thymic diseases, systemic lupus erythematosus);
10. Subjects with positive serological virology tests (HBsAg, HCV antibody, HIV antibody, Treponema pallidum antibody); however, hepatitis B virus carriers, stable hepatitis B patients after drug treatment (DNA titer ≤500 IU/mL or copy number <1000 copies/mL), and cured hepatitis C patients (HCV RNA negative) may be enrolled after being deemed eligible by the investigator;
11. Subjects allergic to human albumin, anesthetic drugs, or any of their components;
12. Subjects who have participated in any other clinical trial within 3 months prior to screening;
13. Subjects who cannot tolerate bronchoscopy (including but not limited to the following conditions: active massive hemoptysis; severe hypertension and arrhythmia; myocardial infarction within 4-6 weeks prior to screening or history of unstable angina; severe cardiopulmonary dysfunction; uncorrectable bleeding tendency (platelet count <60×109/L), such as severe coagulation disorders, uremia, and severe pulmonary hypertension; severe superior vena cava obstruction syndrome; suspected aortic aneurysm; multiple pulmonary bullae; extreme systemic exhaustion);
14. Subjects deemed by the investigator to be at high risk for general/local anesthesia;
15. Pregnant or lactating women, or those with a positive β-human chorionic gonadotropin (β-HCG) test during screening, or those unable or unwilling to adopt effective non-pharmacological contraceptive measures during the study and for 6 months after study completion;
16. Other circumstances deemed by the investigator as unsuitable for participation in this trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Tolerance of patients with idiopathic fibrosis to human umbilical cord mesenchymal stem cell injection | From the first administration to 4 weeks after administration
  Incidence and severity of adverse events according to CTCAE5.0
Dose exploration of patients with idiopathic fibrosis to human umbilical cord mesenchymal stem cell injection | From the first administration to 4 weeks after administration
  The maximum tolerable dose (MTD) of a single administration depends on whether dose limiting toxicity (DLT) occurs within 4 weeks after the first administration, for example (1) Hematological toxicity of grade 3 and above caused by the treatment of human umbilical cord mesenchymal stem cell injection,
  （2） There are grade 3 and above non hematological toxic reactions caused by the treatment of human umbilical cord mesenchymal stem cell injection, except for the following cases, (3) Any other toxicity related to cell therapy that is higher than the baseline level is judged as clinically significant and / or unacceptable by the investigator and the sponsor, (4) There are acute exacerbations and serious adverse events (SAE) of IPF related to the treatment of human umbilical cord mesenchymal stem cell injection (which may be related, likely to be related and definitely related)

SECONDARY OUTCOMES:
Preliminary efficacy evaluation | The 4th, 12th, 24th and 48th week after administration
  Changes from baseline in St. George's respiratory questionnaire SGRQ, dyspnea score, cough score and 6-minute walk test (grade and distance)in the treatment of idiopathic pulmonary fibrosis (IPF), and to recommend the appropriate dose of cell therapy for subsequent clinical studies
Preliminary efficacy evaluation | The 4th, 12th, 24th and 48th week after administration
  Changes in lung function (FVC, DLCO sb) compared with baseline

OTHER OUTCOMES:
Preliminary efficacy evaluation | The 4th, 12th, 24th and 48th week after administration
  Changes in abnormal values of routine safety tests (blood routine, urine routine, blood biochemistry, 12 lead ECG, etc.) compared with baseline
Preliminary efficacy evaluation | The 12th, 24th and 48th week after administration
  Changes in chest HRCT scores from baseline
Preliminary efficacy evaluation | The 12th, 24th and 48th week after administration
  Changes of lung tumor markers from baseline
Preliminary efficacy evaluation | Within 48 weeks after administration
  Frequency and severity of acute exacerbations of IPF
Immunogenicity of human umbilical cord mesenchymal stem cells | The 1st and 4th weeks after administration
  Changes of specific immunoglobulin G (IgG) from baseline
Immunogenicity of human umbilical cord mesenchymal stem cells | The 1st and 4th weeks after administration
  Cytokines (TNF- α、 IFN- γ、 Changes of IL-2, IL-4, IL-5 and IL-6) from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Glassberg MK, Minkiewicz J, Toonkel RL, Simonet ES, Rubio GA, DiFede D, Shafazand S, Khan A, Pujol MV, LaRussa VF, Lancaster LH, Rosen GD, Fishman J, Mageto YN, Mendizabal A, Hare JM. Allogeneic Human Mesenchymal Stem Cells in Patients With Idiopathic Pulmonary Fibrosis via Intravenous Delivery (AETHER): A Phase I Safety Clinical Trial. Chest. 2017 May;151(5):971-981. doi: 10.1016/j.chest.2016.10.061. Epub 2016 Nov 24. PMID 27890713
- [Background] Tzouvelekis A, Paspaliaris V, Koliakos G, Ntolios P, Bouros E, Oikonomou A, Zissimopoulos A, Boussios N, Dardzinski B, Gritzalis D, Antoniadis A, Froudarakis M, Kolios G, Bouros D. A prospective, non-randomized, no placebo-controlled, phase Ib clinical trial to study the safety of the adipose derived stromal cells-stromal vascular fraction in idiopathic pulmonary fibrosis. J Transl Med. 2013 Jul 15;11:171. doi: 10.1186/1479-5876-11-171. PMID 23855653
- [Background] Chambers DC, Enever D, Ilic N, Sparks L, Whitelaw K, Ayres J, Yerkovich ST, Khalil D, Atkinson KM, Hopkins PM. A phase 1b study of placenta-derived mesenchymal stromal cells in patients with idiopathic pulmonary fibrosis. Respirology. 2014 Oct;19(7):1013-8. doi: 10.1111/resp.12343. Epub 2014 Jul 9. PMID 25039426
- [Background] Moodley Y, Atienza D, Manuelpillai U, Samuel CS, Tchongue J, Ilancheran S, Boyd R, Trounson A. Human umbilical cord mesenchymal stem cells reduce fibrosis of bleomycin-induced lung injury. Am J Pathol. 2009 Jul;175(1):303-13. doi: 10.2353/ajpath.2009.080629. Epub 2009 Jun 4. PMID 19497992
- [Background] Hass R, Kasper C, Bohm S, Jacobs R. Different populations and sources of human mesenchymal stem cells (MSC): A comparison of adult and neonatal tissue-derived MSC. Cell Commun Signal. 2011 May 14;9:12. doi: 10.1186/1478-811X-9-12. PMID 21569606
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066